CLINICAL TRIAL: NCT06069076
Title: Diagnostic Value of Serum Cathepsin S and Chromogranin A in Diabetic Kidney Disease
Brief Title: Diagnostic Value of Serum Cathepsin S and Chromogranin A in DKD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Z A Kamel, principal investigator, Assiut University
Other Study IDs: Diabetic kidney disease
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cathepsin S and chromogranin A — Diagnostic value of serum Cathepsin S and Chromogranin A

SUMMARY:
1. Evulate the diagnostic value of serum cathepsin S and chromogranin A for Diabetic kidney disease.
2. To correlate the levels of serum Cathepsin S and chromogranin A with HbA1c and eGFR in type 2 diabetic patients based on urinary Albumin- Creatinine Ratio.

DETAILED DESCRIPTION:
Diabetic nephropathy (DN) is a common and serious complication of diabetes and has been shown to be a major cause of end-stage renal disease (ESRD), requiring costly renal replacement therapy in the form of dialysis or transplantation .

It is appreciated that up to 40% of patients with type 1 and type 2 diabetes mellitus (DM) present DN . Early detection and appropriate treatment are essential to prevent disability and death.

Cathepsin S (Cat-S) was a secreted cysteine proteolytic enzyme that is mainly expressed in macrophages. Macrophages undergoing chemotaxis adhere to the basement membrane of blood vessels and secrete Cat-S, and the secreted Cat-S was involved in hydrolysis of elastin, laminin, collagen and other extracellular matrix components, causing vascular damage .

So, Cathepsin S(Cat-S), a novel non-invasive diagnostic marker mediates vascular endothelial dysfunction.

In recent years, studies have shown that up regulation of Cat-S was associated with the development of IgA nephropathy, lupus nephritis, insulin resistance, diabetes and other renal diseases.

Chromogranin A (CgA) is the main member of the chromogranin family and is an acidic glycoprotein consisting of 439 amino acids with an approximate molecular mass of 48 kDa. CgA is used as a diagnostic marker of neuroendocrine tumors(6). The kidney is the main site for the removal of CgA, and it is retained in serum with declining renal function. In patients with renal failure, serum CgA increases much more than creatinine and the other studied low-MW proteins.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as type 2 Diabetes mellitus
* Patients with T2DM with normoalbuminuria , microalbuminuria and macroalbuminuria.

Exclusion Criteria:

* Renal impairment of other Known origin,
* Type 1 D,
* Hepatic disease,
* Heart failure,
* Thyroid disorders,
* Autoimmune disorders,
* Inflammatory condition,
* Malignancy,
* Urinary tract infection,
* Pregnancy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 diabetes mellitus from age 20 years to 80 years
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Evulate the diagnostic value of serum cathepsin S and chromogranin A for Diabetic kidney disease. | Baseline
  Evaluation of the clinical utility of the measurement of the level of Cathepsin S and chromogranin A in type 2 diabetic nephropathy.

SECONDARY OUTCOMES:
correlate the levels of serum Cathepsin S and chromogranin A with HbA1c and eGFR in type 2 diabetic patients based on urinary Albumin- Creatinine Ratio. | Baseline
  Studying the correlation of the levels of serum Cathepsin S and chromogranin A with HbA1c and eGFR in type 2 diabetic patients based on urinary Albumin- Creatinine Ratio.

REFERENCES:
- [Background] Ren X, Wang W, Cao H, Shao F. Diagnostic value of serum cathepsin S in type 2 diabetic kidney disease. Front Endocrinol (Lausanne). 2023 May 25;14:1180338. doi: 10.3389/fendo.2023.1180338. eCollection 2023. PMID 37305031
- [Background] Yu H, Wang H, Su X, Cao A, Yao X, Wang Y, Zhu B, Wang H, Fang J. Serum chromogranin A correlated with albuminuria in diabetic patients and is associated with early diabetic nephropathy. BMC Nephrol. 2022 Jan 21;23(1):41. doi: 10.1186/s12882-022-02667-0. PMID 35062888